CLINICAL TRIAL: NCT05182918
Title: Substance Use and Lifestyle-related Health Problems Among Ageing Patients in OMT and Other SUD Treatment
Brief Title: Substance Use and Lifestyle-related Health Problems in Ageing Patients in OMT Treatment
Acronym: AgeSUD
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Other Study IDs: 813485
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2021-12

CONDITIONS: Substance Use Disorders; Opioid Use Disorder; Tobacco Use; Health, Subjective; Mental Health Impairment
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in OMT and other SUD treatment: Patients in opioid maintenance treatment and other substance use disorder treatment
  Interventions: Other: Substance use disorder treatment

INTERVENTIONS:
Other: Substance use disorder treatment — The study followed a heterogenous sample of patients in opioid maintenance treatment (OMT) and other substance use disorder treatment. The main focus was on health related problems in this cohort, with focus on tobacco use and substance use.

SUMMARY:
The overall aim of the study is to explore substance use, tobacco use and lifestyle-related health problems among ageing patients in Opioid Maintenance Treatment (OMT), and other SUD treatment.

The study will use already collected data from the multi-center, longitudinal, observational NorComt study (Norwegian Cohort of Patients in Opioid Maintenance Treatment and Other Drug Treatment study).

NorComt is the largest longitudinal study of SUD patients in Norway. The data consists of data from OMT and other substance use disorders (SUD) treatment (N=548).

DETAILED DESCRIPTION:
The overall aim of the study is to explore substance use, tobacco use and lifestyle-related health problems among ageing patients in Opioid Maintenance Treatment (OMT), and other SUD treatment.

The study will use already collected data from the multi-center, longitudinal, observational NorComt (Norwegian Cohort of Patients in Opioid Maintenance Treatment and Other Drug Treatment) study.

NorComt is the largest longitudinal study of SUD patients in Norway. The data consists of data from OMT and other substance use disorders (SUD) treatment (N=548).

The present doctoral research degree project is financed by the Southern and Eastern Norway Regional Health Authority, and hosted by Sørlandet hospital in collaboration with the Norwegian Centre for Addiction Research (SERAF).

Ethical approval for analysis of NorComt data and for the planned registry data linkages of NorComt data has been granted by the Norwegian Regional Ethics Committee (REK 2012/1131).

ELIGIBILITY:
Inclusion Criteria:

* Admittance to a substance use disorder treatment facility, either standardized opioid maintenance treatment (OMT) or other substance use disorder treatment (in-patient)

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were included in the study from 21 participating treatment facilities across Norway, 14 were opioid maintenance treatment (OMT) outpatient centers, and 7 were inpatient centers (predominately non-OMT). Apart from an established opioid use disorder diagnosis there are no further criteria for entering OMT treatment, although generally substitution free treatment is recommended as a first option. In-patient SUD treatment represented in the present project typically has a duration of 6-9 months, primarily with non-OMT treatment in therapeutic community-like settings. Some patients would transfer to an outpatient treatment after completing in-patient treatment.
Sampling Method: Non-Probability Sample
Enrollment: 548 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Tobacco use | Approximately one year after admission to treatment (range 11 - 18 months)
  Changes in tobacco use from baseline to follow-up
Substance use | Approximately one year after admission to treatment (range 11 - 18 months)
  Changes in substance use from baseline to follow-up. Excerpts from the European version were used to collect data on substance use. Substance use was scored for the previous 4 weeks on a 6-point response format were 0 corresponded to "No use" and 5 corresponded to "Daily use". 1 year follow-up were compared with baseline values.
Somatic complaints. | Approximately one year after admission to treatment (range 11 - 18 months).
  Changes in somatic complaints from baseline to follow-up. A checklist containing 16 somatic complaints common among chronic drug users, including major organ systems. Responses are provided on a 0 -4 response format, with 0 corresponding to "not at all", 1 "a little", 2 "moderately", 3 "a lot", and 4 "very much".

SECONDARY OUTCOMES:
Mental distress | Approximately one year after admission to treatment (range 11 - 18 months)
  Changes from baseline to post-treatment and follow-up. The Hopkins Symptom Checklist (HSCL) 25-item version was used to measure mental distress. Each of the 25 items was scored on a 5-point scale (0-4). An average score was computed, indicating a global severity index of mental distress (GSI).
QoL (quality of life) | Approximately one year after admission to treatment (range 11 - 18 months)
  Excerpts from the QoL10 will be used to assess QoL. The scale has 10 ordinal items and each item is scored from 1 = very poor up to 5 = very good. The scale is transformed to a decimal scale ranging from 0.1 to 0.9 and averaged, where 0.9 is the best QoL. A normative score in a population sample was 0.7.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clausen, PhD, Principal Investigator — Norwegian Centre for Addiction Research, University of Oslo
Locations (1):
- Addiction Unit - Sørlandet Hospital, Kristiansand, Agder, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data can be shared upon reasonable request

REFERENCES:
- [Derived] Bjornestad ED, Vederhus JK, Clausen T. Change in substance use among patients in opioid maintenance treatment: baseline to 1-year follow-up. Harm Reduct J. 2024 May 24;21(1):101. doi: 10.1186/s12954-024-01005-x. PMID 38790008
- [Derived] Bjornestad ED, Vederhus JK, Clausen T. Change in self-reported somatic symptoms among patients in opioid maintenance treatment from baseline to 1-year follow-up. BMC Psychiatry. 2024 Feb 21;24(1):149. doi: 10.1186/s12888-024-05590-w. PMID 38383345